CLINICAL TRIAL: NCT05732454
Title: A PHASE 2/3, TWO-PART STUDY TO EVALUATE THE EFFICACY AND LONG-TERM SAFETY WITH ORAL ETRASIMOD, 2 MG, ONCE DAILY IN ADULT PARTICIPANTS WITH MODERATE-TO-SEVERE ATOPIC DERMATITIS WITH A HISTORY OF PRIOR SYSTEMIC TREATMENT FAILURE
Brief Title: A Study to Learn About the Study Medicine Etrasimod in Adults With Moderate to Severe Atopic Dermatitis (AD) Who Have Already Tried Treatments Taken by Mouth or by Injection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Per the results of the planned interim analysis, the study met futility criteria for efficacy so the trial was terminated. This decision was made for efficacy reasons only and is not due to any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C5041005; 2022-003361-37 (EudraCT Number); APD334-314 (Other: Alias Study Number)
Record Dates: First submitted 2022-12-22; First posted 2023-02-17 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis, Unspecified; Eczema; Eczema, Atopic
Keywords: Systemic Failure; Oral
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — etrasimod

STUDY DESIGN:
Intervention Model Description: Part 1: Approximately 60 participants with moderate-to-severe AD with a history of prior systemic treatment failure will be randomized (1:1 ratio) in a double blind (DB) manner to receive etrasimod 2 mg or placebo orally, once daily, for 16 weeks. Randomization will be stratified by disease severity as measured by IGA score (3 [moderate AD], 4 [severe AD]) at baseline.
  After DB period, participants may be given the option to continue in an open label extension (OLE) phase whereby they will receive etrasimod 2 mg (tablet) for up to an additional 52 weeks.
  Part 2: Approximately 340 additional participants will be enrolled to receive etrasimod 2 mg orally, once daily, for 52 weeks in an open-label manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PART 1 Double Blind portion (Day 1 through Week 16): all parties are blinded to treatment.
  PART 1 Open Label Extension portion: All parties will be aware participant is taking etrasimod for up to an additional 52 weeks.
  PART 2 Open Label All parties will be aware participant is taking etrasimod for 52 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- etrasimod (Experimental): 2 mg, oral tablet, once daily
  Interventions: Drug: etrasimod
- Placebo (Part 1 DB period only) (Placebo Comparator): Oral sham comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: etrasimod — PART 1 Double Blind one 2 mg tablet once daily for up to 16 weeks PART 1 Open Label Extension one 2 mg tablet once daily for an additional 52 weeks PART 2 Open Label one 2 mg tablet once daily for up 52 weeks
  Other Names: APD334; PF-07915503
  Arms: etrasimod
Drug: Placebo — PART 1 DOUBLE BLIND Placebo - one table daily for up to 16 weeks
  Arms: Placebo (Part 1 DB period only)

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine called etrasimod for the possible treatment of atopic dermatitis (AD), also called eczema, in adults who have already tried AD treatments taken by mouth or by injection that work all over the body. These adults can have moderate to severe AD.

This study is seeking participants who:

* have AD for at least 1 year
* have moderate-to-severe AD
* have tried treatments that work all over the body and saw no effects
* are willing to apply a moisturizer at least once daily during the study

This is a 2-part study that is only selecting about 60 participants for Part 1 as of now. In Part 1, half of the participants will receive etrasimod, a pill to be taken by mouth once daily. The other half will receive a placebo, a pill that looks like etrasimod but has no medicine also taken by mouth once daily. No one will know what treatment the participant is taking. The Sponsor will compare participant experiences of those taking etrasimod to those taking placebo for 16 weeks. This will help determine if the study medicine is safe and effective. After the first 16 weeks, some participants may continue the study knowing they are taking etrasimod for an additional 52 weeks.

Those participating for just the first 16-weeks, will need to visit the study clinic at least 6 times during the study (about every 4 weeks), and will have to come for 2 safety follow up visits at 2nd and 4th week after the last dose of study medicine. People who want to and can continue for an additional 52 weeks will need to visit the study clinic for at least 6 more visits making 12 total visits over 68 weeks followed by 2 safety follow up visits at the 2nd and 4th week after the last dose of study medicine.

In Part 2 of the study, around 340 more participants will be participating. Everyone will receive etrasimod pills once daily for 52 weeks. Participants will need to go to the study clinic at least 9 times after which they will have to go for 2 more safety follow up visits at the 2nd and 4th weeks after the last dose of study medicine.

At every study visit in Part 1 and Part 2, the focus will be on signs and symptoms of AD (like lesions, itch, and pain) as well as general health and overall side effects. Blood samples and vital signs will be taken at every visit. Due to the way the study medicine works, the in-study clinic visit will last at least 4 hours on Day 1 (Part 1 and Part 2) and Week 16 (Part 1).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following key inclusion criteria to be eligible for enrollment into the study:

1. Age 18-80 at screening (or minimum age of consent according to local regulations).

2 Chronic AD (also known as atopic eczema) that was diagnosed at least 1 year prior to Screening and meets Hanifin and Rajka criteria at screening).1 3. Moderate to severe AD:

1. IGA score ≥3 (on the 0 to 4 IGA scale, in which 3 = moderate and 4 = severe) at screening and baseline (Day 1)
2. BSA ≥10% of AD involvement at screening and baseline (Day 1)
3. Eczema Area and Severity Index (EASI) ≥16 at screening and baseline (Day 1) 4. A participant who has failed a prior systemic therapy for AD, ie, refractory, moderate-to-severe AD that is not adequately controlled with other systemic drug products, including biologics, or when use of those therapies is inadvisable.

   5. Willing to apply a topical emollient/moisturizer at least once daily for ≥1 week prior to baseline (Day 1) and willing to maintain consistent (ie, no change in type, frequency, or application) daily application over the course of the study.

   Exclusion Criteria:

   Participants are excluded from the study if any of the following criteria apply:

   Medical Conditions:
   1. Presence of confounding factors:

      * Skin conditions (eg, psoriasis, seborrheic dermatitis) that may interfere with evaluation of AD or assessment of treatment response as deemed by the investigator.
      * Current significant active infection or requiring a treatment for infection that may interfere with the assessment of AD.
   2. Hypersensitivity to etrasimod or any of the excipients.
   3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- United States (44):
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Jared R. Younger, MD (Ophthalmologist), Fountain Valley, California
  - Bryan D. Vo. MD (Pulmonologist), Laguna Hills, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Dr. Carolyn M. Wong, Los Angeles, California
  - Dr. Gerald Markovitz, Los Angeles, California
  - Resolution Advanced Imaging Center, Santa Monica, California
  - Ponce PFT & Medical services, INC [for pulmonology examination], Aventura, Florida
  - Advanced Eye Center: Rodrigo Belalcazar, MD, Hialeah, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Gsi Clinical Research, Margate, Florida
  - Randy Burks, MD, FACS, Margate, Florida
  - D & H National Research Centers, Inc., Miami, Florida
  - Imaging - Advanced Health Imaging, Miami, Florida
  - The Selem Center [Ophthalmologist JOSEPH SELEM], Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Ophthalmology - Dr. Edward Boshnick's Global Vision Rehabilitation Center, Miami, Florida
  - Pulmonology - Miami Pulmonology Specialists, Miami, Florida
  - Pelletier Jesse MD, North Miami Beach, Florida
  - Santos Carlos R MD, North Miami Beach, Florida
  - Tory Sullivan, Md Pa, North Miami Beach, Florida
  - Gateway Radiology, Pinellas Park, Florida
  - Hull & Hull Medical Specialists, Plantation, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - St. Anthonys Hospital, St. Petersburg, Florida
  - USF Health, Tampa, Florida
  - Lung and Sleep Disorder Center, Lathrup Village, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Somerset Opthalmology PC, Troy, Michigan
  - Eye Institute, Tulsa, Oklahoma
  - Pulmonary and Sleep Center of Oklahoma, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - In Vision Optical and Eyecare, Rapid City, South Dakota
  - Eye Care Associates of Arlington, Arlington, Texas
  - Arlington Research Center, Arlington, Texas
  - Texas Pulmonary, Arlington, Texas
  - Alpesh D. Desai, DO PLLC, Houston, Texas
  - Becky Fredrickson, MD [Optometrist/Ophthalmologist], Houston, Texas
  - Rupesh Vakil, MD [Pulmonologist], Houston, Texas
  - Acclaim Dermatology, Sugar Land, Texas
  - Horizon Eye Care and Optical, Sugar Land, Texas
  - Sweetwater Pulmonary Associates, Sugar Land, Texas
- Canada (5):
  - Rejuvenation Dermatology, Edmonton, Alberta
  - CaRe Clinic, Red Deer, Alberta
  - Visique, Québec, Quebec
  - Biron, Québec
  - Alpha Recherche Clinique, Québec
- Czechia (3):
  - Poliklinika VEKTOR Pardubice, Pardubice
  - Pratia Pardubice a.s., Pardubice
  - Fakultní nemocnice v Motole, Prague
- Poland (22):
  - Flosmed, Poznan, Greater Poland Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej Zespół Poradni Specjalistycznych "Termedica", Poznan, Greater Poland Voivodeship
  - Medoculis, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne ,,All - Med'' Badania Kliniczne, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Dietla 19, Krakow, Lesser Poland Voivodeship
  - Artemed Centrum Medyczne, Wroclaw, Lower Silesian Voivodeship
  - Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - Specjalistyczna Praktyka Lekarska Joanna Kalinowska, Wroclaw, Lower Silesian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Michał Silber, Wroclaw, Lower Silesian Voivodeship
  - DERMEDIC Iwona Zdybska, Lublin, Lublin Voivodeship
  - Eyemed, Lublin, Lublin Voivodeship
  - AUGON Gabinet Okulistyczny, Bialystok, Podlaskie Voivodeship
  - Nzoz Specjalistyczny Ośrodek Dermatologiczny "Dermal", Bialystok, Podlaskie Voivodeship
  - Gabinet Alergologiczny IR-med dr n. med. Izabela Roszko-Kirpsza, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Centrum Zdrowia Ochaliczówka, Katowice, Silesian Voivodeship
  - Medicus, Szczecin, West Pomeranian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - Gabinety Lekarskie Rivermed, Poznan
  - Centrum Medyczne Szpital Świętej Rodziny, Lodz, Łódź Voivodeship
  - Dermoklinika - Centrum Medyczne spółka cywilna M. Kierstan, J. Narbutt, A. Lesiak, Lodz, Łódź Voivodeship
  - Ekovivus, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5041005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had 2 parts: Part 1 and Part 2. Part 2 was never initiated; hence no results are reported for it. All results are pertaining to Part 1 in the record. Part 1 of the study had 16-week double-blind (DB) treatment period and then 52-week part 1 open label extension (OLE) treatment period.
Pre-assignment Details: A total of 58 participants with moderate-to-severe atopic dermatitis (AD) were enrolled in Part 1- DB period and out of them 51 continued into the Part 1- OLE period.
Groups:
- DB Etrasimod 2 mg Then OLE Etrasimod 2 mg: Participants were randomized to receive etrasimod 2 milligram (mg) orally once daily for 16 weeks in DB period of Part 1. Eligible participants per investigator's judgement then continued to receive etrasimod 2 mg orally once daily for maximum of another 52 weeks in OLE period of Part 1.
- DB Placebo Then OLE Etrasimod 2 mg: Participants were randomized to receive placebo matched to etrasimod 2 mg orally once daily for 16 weeks in DB period of Part 1. Eligible participants per investigator's judgement then received etrasimod 2 mg orally once daily for maximum of another 52 weeks in OLE period of Part 1.
Period: Part 1: DB Period
Arm/Group | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg | DB Placebo Then OLE Etrasimod 2 mg
Started | 30 | 28
Completed | 27 | 25
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Period: Part 1: OLE Period
Arm/Group | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg | DB Placebo Then OLE Etrasimod 2 mg
Started | 27 (Participants who entered OLE period upon completion of DB period.) | 24 (Participants who entered OLE period upon completion of DB period.)
Completed | 0 | 0
Not Completed | 27 | 24
Not completed — Study Terminated by Sponsor | 25 | 19
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized to the study irrespective of whether they received any dose of study intervention (i.e., Etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg | DB Placebo Then OLE Etrasimod 2 mg | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (14.78) | 43.4 (18.18) | 41.6 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 9 | 30
  Male | 9 | 19 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 24 | 27 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1, DB Period: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response at Week 16
Description: IGA measured AD severity, based on a 5-point scale (0-4); 0= AD is clear, 1= AD is almost clear, 2= mild AD, 3= moderate AD and 4= severe AD. IGA response was defined as participants achieving IGA 0 (clear) or 1 (almost clear) and a reduction of >=2 points from baseline.
Time Frame: DB Period: Week 16
Population: FAS included all participants who were randomized to the study irrespective of whether they received any dose of study intervention (i.e., etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized. Number of participants in FAS with baseline IGA>=2 was included in this analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- DB Period: Etrasimod 2 mg: Participants who received etrasimod 2 mg orally once daily for 16 weeks in DB period of Part 1.
- DB Period: Placebo: Participants who received placebo matched to etrasimod orally once daily for 16 weeks in DB period of Part 1.
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Percentage of Participants | 3.3 [lower limit 3.28] | 7.1 [lower limit 4.87]
Statistical Analysis 1: Comparison: DB Period: Etrasimod 2 mg vs DB Period: Placebo; Normal approximation adjusting for the stratification factor (disease severity as measured by baseline IGA score 3 [moderate], 4 [severe]) derived from clinical database via Cochran-Mantel-Haenszel (CMH) approach was used; Test type: Superiority; p = 0.5580, Cochran-Mantel-Haenszel; Difference in percentage = -3.76, 95% CI 2-sided [-16.36 to 8.83]

2. Secondary Outcome: Part 1, DB Period: Percentage of Participants Who Achieved >=75% Reduction From Baseline in Eczema Area and Severity Index (EASI) Score (EASI-75) at Week 16
Description: EASI-75 response was defined as a 75% reduction or greater in EASI score from Baseline to Week 16. EASI quantified severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema [E], induration/papulation [I], excoriation [Ex] and lichenification [L]) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; h = head and neck; u = upper limbs; t = trunk; l = lower limbs.
Time Frame: DB Period: Week 16
Population: FAS included all participants who were randomized to the study irrespective of whether they received any dose of study intervention (i.e., etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Percentage of Participants | 23.3 [lower limit 7.72] | 14.3 [lower limit 6.61]
Statistical Analysis 1: Comparison: DB Period: Etrasimod 2 mg vs DB Period: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3685, Cochran-Mantel-Haenszel; Difference in percentage = 9.07, 95% CI 2-sided [-10.70 to 28.85]

3. Secondary Outcome: Part 1, DB Period: Percent Change From Baseline in EASI Score at Week 16
Description: EASI quantified severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema [E], induration/papulation [I], excoriation [Ex] and lichenification [L]) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; h = head and neck; u = upper limbs; t = trunk; l = lower limbs.
Time Frame: DB Period: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Percent change | -53.87 (9.007) | -24.65 (9.533)
Statistical Analysis 1: Comparison: DB Period: Etrasimod 2 mg vs DB Period: Placebo; Jump-to-Control (JTC) method was used for evaluation. A complete imputed dataset was analyzed using analysis of covariance model including effects of treatment group, actual stratification factor, and baseline value. Multiple results of the treatment comparison were combined using Rubin's rules, reporting the combined treatment difference, its standard error, 95% CI and 2-sided p-value, across the visits; Test type: Superiority; p = 0.0303, Rubin's rule; Difference in Mean = -29.22, 95% CI 2-sided [-55.53 to -2.90]

4. Primary Outcome: Part 1, DB Period: Number of Participants With Treatment Emergent Adverse Events (TEAEs) (All Causality)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: DB Period: From first dose of study drug up to 16 Weeks of treatment
Population: DB period: Safety analysis set included of all participants who were randomized and received at least 1 dose of study drug in DB period.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants | 16 | 8

5. Primary Outcome: Part 1, DB Period: Number of Participants With TEAEs (All Causality) Leading to Study Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: DB Period: From first dose of study drug up to 16 Weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants | 1 | 0

6. Primary Outcome: Part 1, DB Period: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) (All Causality)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to last dose that were absent before treatment or that worsened relative to pretreatment state. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of death); new or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or other medical events judged by investigator.
Time Frame: DB Period: From first dose of study drug up to 16 Weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants | 0 | 0

7. Primary Outcome: Part 1, DB Period: Number of Participants With Treatment Emergent AEs of Special Interest (AESIs) (All Causality)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to last dose that were absent before treatment or that worsened relative to pretreatment state. AESIs included here were cardiovascular events (i.e., bradycardia, Atrioventricular (AV) conduction delay, and hypertension); macular edema, pulmonary events (airflow obstruction or decreased gas exchange); infections (severe infections, opportunistic infections [including progressive multifocal leukoencephalopathy (PML)], Herpes simplex and Herpes zoster); liver injury (liver transaminase elevation and bilirubin elevation); posterior reversible encephalopathy syndrome (PRES) and malignancies.
Time Frame: DB Period: From first dose of study drug up to 16 Weeks of treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants | 2 | 1

8. Primary Outcome: Part 1, DB Period: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory assessments included hematology, clinical chemistry, urinalysis, other parameters and reflex tests. Number of participants with abnormalities in any of laboratory parameters is reported.
Time Frame: DB Period: From first dose of study drug up to 16 Weeks of treatment
Population: DB period: Safety analysis set included of all participants who were randomized and received at least 1 dose of study drug in DB period. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 29 | 27
Participants | 22 | 13

9. Primary Outcome: Part 1, DB Period: Number of Participants With Markedly Abnormal 12-Lead Electrocardiogram Measurements and AV Blocks
Description: Standard 12-lead ECGs utilizing limb leads were used to measure PR interval, QT interval, QTc corrected using Fridericia's formula (QTcF), and QRS complex. Number of participants with non-zero ECG abnormalities and AV blocks are reported in this outcome measure.
Time Frame: DB Period: Pre-dose and 4 hours (hrs) post-dose on Day 1/Week 0; Pre-dose and 4 hrs post-dose on Day 113/Week 16
Population: DB period: Safety analysis set included of all participants who were randomized and received at least 1 dose of study drug in DB period. Here, "Number Analyzed"= number of participants evaluable for specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants
  Pre-dose/Day 1: AV conduction: First-degree AV Block | 1 | 0
  4 hrs post-dose/Day 1: QTCF (msec), single beat:>= 450 (male) or >= 470 (female) | 1 | 0
  4 hrs post-dose/Day 1: Change From Baseline (CFB) in QT: >30 msec increase | 9 | 0
  4 hrs post-dose/Day 1: AV conduction: First degree AV Block | 3 | 0
  Pre-dose/Week 16: CFB in QT: >30 msec increase: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: CFB in QT: >30 msec increase | 1 | 0
  Pre-dose/Week 16: CFB in QT: >60 msec increase: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: CFB in QT: >60 msec increase | 1 | 0
  Pre-dose/Week 16: CFB in QTcF: >30 msec increase: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: CFB in QTcF: >30 msec increase | 2 | 0
  4 hrs post-dose/Week 16: CFB in QTcF: >30 msec increase: number analyzed (Participants) | 25 | 24
  4 hrs post-dose/Week 16: CFB in QTcF: >30 msec increase | 2 | 0
  4 hrs post-dose/Week 16: CFB in QT: >30 msec increase: number analyzed (Participants) | 25 | 24
  4 hrs post-dose/Week 16: CFB in QT: >30 msec increase | 2 | 0
  4 hrs post-dose/Week 16: AV conduction: First degree AV Block: number analyzed (Participants) | 25 | 24
  4 hrs post-dose/Week 16: AV conduction: First degree AV Block | 2 | 0

10. Primary Outcome: Part 1, DB Period: Number of Participants With Markedly Abnormal Vital Sign
Description: Vital signs evaluation included systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate. Number of participants with non-zero vital signs abnormalities are reported in this outcome measure.
Time Frame: DB Period: Pre-dose and 1, 2, 3, 4 hours (hrs) post-dose on Day 1/Week 0; Day 29/Week 4; Day 57/Week 8; Day 85/Week 12; Pre-dose and 1, 2, 3, 4, 5 and 6 hrs post-dose on Day 113/Week 16
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo
Number analyzed (Participants) | 30 | 28
Participants
  Pre-dose/Day 1: DBP >90 mmHg | 0 | 1
  Pre-dose/Day 1: Pulse rate: <60 bpm | 1 | 3
  Pre-dose/Day 1: Pulse rate >100 bpm | 1 | 0
  1 hr post-dose/Day 1: SBP: Change >=30 mmHg decrease | 0 | 1
  1 hr post-dose/Day 1: DBP >90 mmHg | 2 | 2
  1 hr post-dose/Day 1: Pulse rate: <50 bpm | 1 | 0
  1 hr post-dose/Day 1: Pulse rate: <60 bpm | 7 | 3
  2 hrs post-dose/Day 1: SBP: >150 mmHg | 0 | 2
  2 hrs post-dose/Day 1: DBP >90 mmHg | 0 | 1
  2 hrs post-dose/Day 1: Pulse rate: <60 bpm | 12 | 5
  3 hrs post-dose/Day 1:SBP >150 mmHg | 0 | 1
  3 hrs post-dose/Day 1: SBP: Change>=30 mmHg decrease | 1 | 0
  3 hrs post-dose/Day 1: DBP:>90 mmHg | 0 | 1
  3 hrs post-dose/Day 1: DBP: Change>=20 mmHg decrease | 2 | 0
  3 hrs post-dose/Day 1: Pulse rate: <60 bpm | 11 | 6
  4 hrs post-dose/Day 1: DBP: >90 mmHg | 1 | 1
  4 hrs post-dose/Day 1: Pulse rate: <60 bpm | 10 | 5
  4 hrs post-dose/Day 1: Pulse rate: >100 bpm | 1 | 0
  Week 4: DBP:>90 mmHg: number analyzed (Participants) | 29 | 27
  Week 4: DBP:>90 mmHg | 2 | 3
  Week 4: Pulse rate: <60 bpm: number analyzed (Participants) | 28 | 27
  Week 4: Pulse rate: <60 bpm | 2 | 1
  Week 4: Pulse rate: >100 bpm: number analyzed (Participants) | 28 | 27
  Week 4: Pulse rate: >100 bpm | 1 | 0
  Week 8: SBP: >150 mmHg: number analyzed (Participants) | 28 | 25
  Week 8: SBP: >150 mmHg | 0 | 1
  Week 8: DBP:>90 mmHg: number analyzed (Participants) | 28 | 25
  Week 8: DBP:>90 mmHg | 3 | 3
  Week 8: DBP: Change >=20 mmHg decrease: number analyzed (Participants) | 28 | 25
  Week 8: DBP: Change >=20 mmHg decrease | 0 | 1
  Week 8: Pulse rate: <60 bpm: number analyzed (Participants) | 28 | 25
  Week 8: Pulse rate: <60 bpm | 3 | 1
  Week 12: SBP: >150 mmHg: number analyzed (Participants) | 27 | 25
  Week 12: SBP: >150 mmHg | 0 | 1
  Week 12: DBP:>90 mmHg: number analyzed (Participants) | 27 | 25
  Week 12: DBP:>90 mmHg | 1 | 3
  Week 12: Pulse rate: <60 bpm: number analyzed (Participants) | 27 | 25
  Week 12: Pulse rate: <60 bpm | 1 | 0
  Week 12: Pulse rate: >100 bpm: number analyzed (Participants) | 27 | 25
  Week 12: Pulse rate: >100 bpm | 0 | 2
  Pre-dose/Week 16: SBP: >150 mmHg: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: SBP: >150 mmHg | 0 | 1
  Pre-dose/Week 16: DBP: >90 mmHg: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: DBP: >90 mmHg | 2 | 0
  Pre-dose/Week 16: Pulse rate: <60 bpm: number analyzed (Participants) | 26 | 24
  Pre-dose/Week 16: Pulse rate: <60 bpm | 2 | 2
  1 hr post dose/Week 16: SBP: >150 mmHg: number analyzed (Participants) | 26 | 24
  1 hr post dose/Week 16: SBP: >150 mmHg | 0 | 1
  1 hr post-dose/Week 16: SBP: Change >=30 mmHg decrease: number analyzed (Participants) | 26 | 24
  1 hr post-dose/Week 16: SBP: Change >=30 mmHg decrease | 0 | 1
  1 hr post dose/Week 16: DBP: >90 mmHg: number analyzed (Participants) | 26 | 24
  1 hr post dose/Week 16: DBP: >90 mmHg | 2 | 1
  1 hr post dose/Week 16: Pulse rate: <50 bpm: number analyzed (Participants) | 26 | 24
  1 hr post dose/Week 16: Pulse rate: <50 bpm | 1 | 1
  1 hr post dose/Week 16: Pulse rate: <60 bpm: number analyzed (Participants) | 26 | 24
  1 hr post dose/Week 16: Pulse rate: <60 bpm | 3 | 4
  2 hrs post dose/Week 16: SBP: >150 mmHg: number analyzed (Participants) | 26 | 24
  2 hrs post dose/Week 16: SBP: >150 mmHg | 0 | 1
  2 hrs post-dose/Week 16: SBP: Change >=30 mmHg decrease: number analyzed (Participants) | 26 | 24
  2 hrs post-dose/Week 16: SBP: Change >=30 mmHg decrease | 0 | 2
  2 hrs post dose/Week 16: DBP: >90 mmHg: number analyzed (Participants) | 26 | 24
  2 hrs post dose/Week 16: DBP: >90 mmHg | 2 | 2
  2 hrs post dose/Week 16: Pulse rate: <50 bpm: number analyzed (Participants) | 26 | 24
  2 hrs post dose/Week 16: Pulse rate: <50 bpm | 0 | 1
  2 hrs post dose/Week 16: Pulse rate: <60 bpm: number analyzed (Participants) | 26 | 24
  2 hrs post dose/Week 16: Pulse rate: <60 bpm | 3 | 10
  3 hrs post dose/Week 16:DBP: >90 mmHg: number analyzed (Participants) | 26 | 24
  3 hrs post dose/Week 16:DBP: >90 mmHg | 2 | 0
  3 hrs post dose/Week 16: Pulse rate: <50 bpm: number analyzed (Participants) | 26 | 24
  3 hrs post dose/Week 16: Pulse rate: <50 bpm | 0 | 1
  3 hrs post dose/Week 16: Pulse rate: <60 bpm: number analyzed (Participants) | 26 | 24
  3 hrs post dose/Week 16: Pulse rate: <60 bpm | 3 | 9
  4 hrs post dose/Week 16: SBP: >150 mmHg: number analyzed (Participants) | 26 | 24
  4 hrs post dose/Week 16: SBP: >150 mmHg | 0 | 1
  4 hrs post dose/Week 16: DBP:>90 mmHg: number analyzed (Participants) | 26 | 24
  4 hrs post dose/Week 16: DBP:>90 mmHg | 2 | 0
  4 hrs post-dose/Week 16: DBP: Change >=20 mmHg decrease: number analyzed (Participants) | 26 | 24
  4 hrs post-dose/Week 16: DBP: Change >=20 mmHg decrease | 0 | 1
  4 hrs post dose/Week 16: Pulse rate: <50 bpm: number analyzed (Participants) | 26 | 24
  4 hrs post dose/Week 16: Pulse rate: <50 bpm | 0 | 1
  4 hrs post dose/Week 16: Pulse rate:<60 bpm: number analyzed (Participants) | 26 | 24
  4 hrs post dose/Week 16: Pulse rate:<60 bpm | 1 | 6
  5 hrs post dose/Week 16:Pulse rate:<50 bpm: number analyzed (Participants) | 0 | 1
  5 hrs post dose/Week 16:Pulse rate:<50 bpm | 0 | 1
  5 hrs post dose/Week 16:Pulse rate:<60 bpm: number analyzed (Participants) | 0 | 1
  5 hrs post dose/Week 16:Pulse rate:<60 bpm | 0 | 1
  6 hrs post dose/Week 16:Pulse rate:<50 bpm: number analyzed (Participants) | 0 | 1
  6 hrs post dose/Week 16:Pulse rate:<50 bpm | 0 | 1
  6 hrs post dose/Week 16: Pulse rate:<60 bpm: number analyzed (Participants) | 0 | 1
  6 hrs post dose/Week 16: Pulse rate:<60 bpm | 0 | 1

11. Primary Outcome: Part 1, OLE Period: Number of Participants With TEAEs (All Causality)
Description: as for outcome 5
Time Frame: OLE Period: First dose of study drug in OLE period up to 4 weeks after last dose in OLE period (up to maximum of 56 Weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention (i.e., Etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period): Participants who received etrasimod 2 mg in DB period and then continued to receive etrasimod 2 mg orally once daily in OLE period for maximum of another 52 weeks.
- OLE Period: Etrasimod 2 mg (Placebo in DB Period): Participants who received placebo matched to etrasimod in DB period and then received etrasimod 2 mg orally once daily in OLE period for maximum of another 52 weeks.
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 30 | 28
Participants | 9 | 5

12. Primary Outcome: Part 1, OLE Period: Number of Participants With Treatment Emergent AEs (All Causality) Leading to Study Treatment Discontinuation
Description: as for outcome 5
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 30 | 28
Participants | 0 | 1

13. Primary Outcome: Part 1, OLE Period: Number of Participants With Treatment Emergent SAEs (All Causality)
Description: as for outcome 6
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 30 | 28
Participants | 1 | 0

14. Primary Outcome: Part 1, OLE Period: Number of Participants With Treatment Emergent AESIs (All Causality)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to last dose that were absent before treatment or that worsened relative to pretreatment state. AESIs included here were cardiovascular events (i.e., bradycardia, AV conduction delay, and hypertension); macular edema, pulmonary events (airflow obstruction or decreased gas exchange); infections (severe infections, opportunistic infections [including PML], Herpes simplex and Herpes zoster); liver injury (liver transaminase elevation and/or bilirubin elevation); PRES and malignancies.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 30 | 28
Participants | 1 | 0

15. Primary Outcome: Part 1, OLE Period: Number of Participants With Laboratory Test Abnormalities
Description: as for outcome 8
Time Frame: as for outcome 11
Population: Safety analysis set included all participants who received at least 1 dose of study intervention (i.e., Etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 28 | 25
Participants | 20 | 18

16. Primary Outcome: Part 1, OLE Period: Number of Participants With Markedly Abnormal 12-Lead Electrocardiogram Measurements and AV Blocks
Description: Standard 12-lead ECGs utilizing limb leads were used to measure PR interval, QT interval, QTcF, and QRS complex. Number of participants with non-zero ECG abnormalities and AV blocks are reported in this outcome measure.
Time Frame: OLE Period: Day 169/Week 24
Population: Safety analysis set included all participants who received at least 1 dose of study intervention (i.e., Etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for the specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 14 | 11
Participants
  Week 24: QTCF (msec), single beat:>= 450 (male) or >= 470 (female) | 1 | 0
  Week 24: CFB in QTcF: >30 sec increase | 1 | 0
  Week 24: CFB in QT: >30 msec increase | 2 | 0
  Week 24: CFB in QT: >60 msec increase | 1 | 0

17. Primary Outcome: Part 1, OLE Period: Number of Participants With Markedly Abnormal Vital Sign
Description: Vital signs evaluation included SBP, DBP, pulse rate. Number of participants with non-zero vital signs abnormalities are reported in this outcome measure.
Time Frame: OLE Period: Day 141/Week 20; Day 169/Week 24; Day 281/Week 40; Follow Up 1; Follow Up 2
Population: Safety analysis set included all participants who received at least 1 dose of study intervention (i.e., Etrasimod or placebo). Participants were analyzed in the treatment groups as they were randomized. "Number Analyzed"=participants evaluable for specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period)
Number analyzed (Participants) | 26 | 23
Participants
  Week 20: SBP: >150 mmHg | 1 | 1
  Week 20: SBP: Change:>=30 mmHg decrease | 0 | 1
  Week 20: DBP: >90 mmHg | 2 | 1
  Week 20: Pulse rate: <60 bpm | 1 | 0
  Week 24: SBP: >150 mmHg: number analyzed (Participants) | 25 | 21
  Week 24: SBP: >150 mmHg | 0 | 1
  Week 24: SBP: Change:>=30 mmHg decrease: number analyzed (Participants) | 25 | 21
  Week 24: SBP: Change:>=30 mmHg decrease | 0 | 1
  Week 24: DBP: >90 mmHg: number analyzed (Participants) | 25 | 21
  Week 24: DBP: >90 mmHg | 1 | 1
  Week 24: DBP: Change>=20 mmHg decrease: number analyzed (Participants) | 25 | 21
  Week 24: DBP: Change>=20 mmHg decrease | 0 | 1
  Week 24: Pulse rate: <60 bpm: number analyzed (Participants) | 25 | 21
  Week 24: Pulse rate: <60 bpm | 1 | 1
  Week 32: DBP: >90 mmHg: number analyzed (Participants) | 11 | 9
  Week 32: DBP: >90 mmHg | 1 | 0
  Week 40: DBP: >90 mmHg: number analyzed (Participants) | 4 | 3
  Week 40: DBP: >90 mmHg | 1 | 0
  Follow-up 1: DBP: >90 mmHg: number analyzed (Participants) | 21 | 18
  Follow-up 1: DBP: >90 mmHg | 2 | 0
  Follow-up 1: Pulse rate: <60 bpm: number analyzed (Participants) | 21 | 18
  Follow-up 1: Pulse rate: <60 bpm | 1 | 2
  Follow-up 2: DBP: >90 mmHg: number analyzed (Participants) | 21 | 19
  Follow-up 2: DBP: >90 mmHg | 2 | 0
  Follow-up 2: Pulse rate: <60 bpm: number analyzed (Participants) | 21 | 19
  Follow-up 2: Pulse rate: <60 bpm | 1 | 2

ADVERSE EVENTS:
Time Frame: Part 1, DB Period: Day 1 to Week 16; Part 1, OLE Period: Week 20 to Week 68; Part 1, DB +OLE Period: Day 1 to Week 68
Description: The same all-causality treatment-emergent event may appear as both SAE & non-SAE.However, what is presented are distinct events.An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious & non-serious event during study. Safety analysis set was evaluated.
Groups:
- OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period): Participants who received etrasimod 2 mg in DB period, received etrasimod 2 mg orally once daily in OLE period for maximum of another 52 weeks.
- OLE Period: Etrasimod 2 mg (Placebo in DB Period): Participants who received placebo matched to etrasimod in DB period, received etrasimod 2 mg orally once daily in OLE period for maximum of another 52 weeks.
Arm/Group | DB Period: Etrasimod 2 mg | DB Period: Placebo | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) | OLE Period: Etrasimod 2 mg (Placebo in DB Period) | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg | DB Placebo Then OLE Etrasimod 2 mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/30 | 0/28 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 1/30 | 0/28 | 1/30 | 0/28
Other Adverse Events (participants affected / at risk) | 6/30 | 4/28 | 4/30 | 1/28 | 9/30 | 5/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Etrasimod 2 mg (N=30) | DB Period: Placebo (N=28) | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) (N=30) | OLE Period: Etrasimod 2 mg (Placebo in DB Period) (N=28) | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg (N=30) | DB Placebo Then OLE Etrasimod 2 mg (N=28)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Etrasimod 2 mg (N=30) | DB Period: Placebo (N=28) | OLE Period: Etrasimod 2 mg (Etrasimod 2 mg in DB Period) (N=30) | OLE Period: Etrasimod 2 mg (Placebo in DB Period) (N=28) | DB Etrasimod 2 mg Then OLE Etrasimod 2 mg (N=30) | DB Placebo Then OLE Etrasimod 2 mg (N=28)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (5) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT05732454/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT05732454/SAP_001.pdf